CLINICAL TRIAL: NCT07199699
Title: The Safety and Efficacy of Subxiphoid Minimally Invasive Resection of Giant Mediastinal Teratoma Assisted by Double Sternal Elevation
Brief Title: Subxiphoid VATS for Giant Mediastinal Teratoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiang Fan, Chief surgeon, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20250612051346797
Record Dates: First submitted 2025-08-24; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Teratomas; Mediastinal ( Chest) Masses; VATS
MeSH Terms: conditions — Teratoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subxiphoid Minimally Invasive Resection Assisted by Double Sternal Elevation (Experimental)
  Interventions: Procedure: Subxiphoid Minimally Invasive Resection of Giant Mediastinal Teratoma Assisted by Double Sternal Elevation

INTERVENTIONS:
Procedure: Subxiphoid Minimally Invasive Resection of Giant Mediastinal Teratoma Assisted by Double Sternal Elevation — All patients underwent minimally invasive mediastinal tumor resection using a double hook technique via the subxiphoid approach. The procedure was as follows: A 3-4 cm longitudinal incision was made below the xiphoid, and subcutaneous tissue was dissected to reach the anterior rectus sheath. The retroxiphoid space was bluntly dissected, and a thoracoscopic lens was inserted. A double-retractor system was placed in the subxiphoid and suprasternal regions, and retractor height was adjusted to aid in separating tumor adhesions from residual thymic tissue. Blunt dissection was used to separate the tumor from the innominate vein and phrenic nerve. After full tumor mobilization, it was placed into a sterile specimen bag and removed through the incision. The surgical area was rinsed and a mediastinal drainage tube was inserted, and the incision was closed layer by layer.

SUMMARY:
For giant mediastinal teratomas, the only treatment option available is usually open-chest surgery, which causes significant trauma, leads to obvious postoperative pain and may result in long-term complications such as chest wall deformity. Currently, we have developed a new treatment method. We use a double retractor system to pull the upper and lower ends of the sternum, lifting it to obtain sufficient surgical space behind the sternum. This enables us to perform minimally invasive tumor resection through the subxiphoid approach with thoracoscopy. The advantages of this method include reduced surgical trauma and postoperative pain, shortened hospital stay, and improved cosmetic effect

ELIGIBILITY:
Inclusion Criteria:

* Age: 10 - 70 years old, gender unrestricted; Preoperative enhanced CT or MRI confirms anterior mediastinal mass with the maximum diameter ≥ 7 cm; Intraoperative frozen section pathology confirms teratoma (mature or immature type); American Society of Anesthesiologists (ASA) classification grade I - III, with acceptable cardiopulmonary function for single-lung ventilation; No severe thoracic deformity or severe adhesion in the posterior mediastinum (assessed by preoperative imaging); Patients voluntarily sign the informed consent form, understanding the purpose and potential risks of the study.

Exclusion Criteria:

* Tumors invading major blood vessels (such as the innominate vein, superior vena cava, or aorta) or the pericardium require combined vascular/pericardial resection and reconstruction; Tumors crossing the midline and encasing the trachea or esophagus require multidisciplinary joint surgery; Previous mediastinal surgery or radiotherapy history, leading to local anatomical structure disorder; Coagulation dysfunction (INR > 1.5 or platelet count < 50×10⁹/L); Severe immune deficiency (such as HIV infection, long-term glucocorticoid treatment); Pregnant or lactating women; Concurrent other malignant tumors (metastatic lesions need to be excluded); Severe cardiopulmonary diseases (such as COPD GOLD Ⅲ-Ⅳ grade, NYHA cardiac function Ⅲ-Ⅳ grade); Mental illness or cognitive impairment that cannot cooperate with postoperative follow-up; Participated in other clinical trials that may interfere with the results of this study.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of intraoperative and postoperative complications | From the start of the surgery to 30 days after the operation

SECONDARY OUTCOMES:
Complete tumor resection rate | From the start of the surgery to two weeks after the operation
Postoperative function | From the start of the surgery to one month after the operation
  The width of the incision scar (mm) and the Vancouver Scar Scale (VSS, 0-15 points) one month after the operation.
Postoperative Quality of life | From the start of the surgery to six month after the operation
  The EuroQol Five Dimensions Questionnaire (EQ-5D) was used to assess the quality of life after the operation